CLINICAL TRIAL: NCT02820519
Title: Tolerability and Analgesic Efficacy of Loxapine in Patients With Refractory, Chemotherapy-induced Neuropathic Pain
Acronym: LOX2015PILOT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Intolerable high amount of adverse events
Sponsor: University of Witten/Herdecke (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LOX_2015_PILOT; 2014-005440-17 (EudraCT Number)
Record Dates: First submitted 2016-06-14; First posted 2016-07-01 (Estimated); Last update posted 2022-07-01 (Actual); Status verified 2017-08

CONDITIONS: Neuropathic Pain
Keywords: Neuropathic pain; Loxapine; Antipsychotics; Co-Analgesics; Tolerability; Analgesic efficacy
MeSH Terms: conditions — Neuralgia | interventions — Loxapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Loxapine (Experimental): Loxapine Capsules 10 mg Day 1- 14: 10 mg b.i.d Day 15-28: 10 mg t.i.d Day 29-42: 20 mg b.i.d. Day 43-56: 20 mg t.i.d. Dosages will be escalated according to analgesic efficacy and tolerability.
  Interventions: Drug: Loxapine

INTERVENTIONS:
Drug: Loxapine — Loxapine dose escalation according to tolerability and analgesic efficacy
  Other Names: Loxapine Succinate

SUMMARY:
Loxapine is an antipsychotic drug approved for the treatment of schizophrenia in several countries including the United States. In animal studies in mice, loxapine reduced neuropathic pain. Hence, in a proof-of-principle and dose-escalating study the tolerability and analgesic efficacy of loxapine will be evaluated in patients with neuropathic pain.

DETAILED DESCRIPTION:
In this dose-escalating study, 12 patients with refractory, chemotherapy-induced neuropathic pain (including mixed pain) will receive loxapine during four 14-days treatment episodes. The dosage for episode 1 (Days 1-14) will be 10 mg b.i.d., dosages for episodes 2, 3, and 4 will be defined by taking into account tolerability and analgesic efficacy of the former episode. In case of an acceptable tolerability and if a clinically relevant analgesic efficacy is not reached, loxapine dosage will be increased (2nd Episode 10 mg t.i.d, 3rd Episode 20 mg b.i.d., 4th episode 20 mg t.i.d.). In case of an acceptable tolerability and if a clinically relevant analgesic efficacy is reached, loxapine dosage will not be changed. If clinically relevant (serious) adverse events ((S)AEs) occur, loxapine dosage will be reduced or the treatment will be interrupted or stopped irrespective of the analgesic efficacy. A clinically relevant pain reduction / analgesic efficacy is defined by an at least 30% decrease or an absolute decrease of two scale units compared to baseline using 11-point numeric pain rating scale. Patients will receive loxapine as add-on treatment to their usual (analgesic) care.

ELIGIBILITY:
Inclusion Criteria:

* Primarily chemotherapy-induced neuropathic pain (including mixed pain) for at least 3 months refractory to at least one analgesic compound
* Neuropathic pain >= 4 (11-point numeric pain scale) at screening visit (including mixed pain)
* Age >= 18 years
* Body weight between 50 and 150 kg
* Given written informed consent

Exclusion Criteria:

* Participation in other interventional clinical studies (currently or within the last 3 months)
* Parkinson's disease, movement disorders (extrapyramidal signs and symptoms) associated with antipsychotics, neuroleptic malignant syndrome, other syndromes associated with antipsychotics
* Severe hypotension with a syncope in history, glaucoma, urinary retention, epilepsy or other seizure disorders in history, severe dementia, dementia-related psychosis in history, malignancies with a life expectancy of less than 6 months, breast cancer in history, other life-threatening conditions
* Corrected QT interval (QTc) > 460 ms (females) or > 450 ms (males)
* Known alcohol and/or drug abuse
* Concomitant intake of antipsychotics, dopamine agonists (Levodopa, bromocriptine, lisuride, pergolide, ropinirole, cabergoline, pramipexole, apomorphine), alpha-receptor blocking compounds
* Compounds with a strong evidence for a clinically relevant QT interval prolongation or torsade de pointes risk increase
* Strong inhibitors of CYP1A2, CYP2D6, or CYP3A4
* Known CYP2D6 Poor metabolizer status
* Pregnancy or lactation period
* Missing or insufficient contraception in pre- or perimenopausal women
* Close Affiliation with the investigational site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-06-07; Primary Completion 2017-05-04 (Actual); Study Completion 2017-05-04 (Actual)

PRIMARY OUTCOMES:
Loxapine dosage with the lowest incidence of events. | After each of the four 14 days study episodes (Day 15, Day 29, Day 43, Day 57)
  The primary endpoint is defined as the first occurrence of a (serious) adverse event ((S)AE) leading to dose reduction or withdrawal of loxapine ("event"). The loxapine dosage with the lowest incidence of events will be identified.

SECONDARY OUTCOMES:
Number, type, and severity of (serious) adverse events ((S)AEs) | After each of the four 14 days study episodes (Day 15, Day 29, Day 43, Day 57)
  Number, type, and severity of (serious) adverse events ((S)AEs)
Cumulative incidence rates for (S)AE pattern of study participants | After each of the four 14 days study episodes (Day 15, Day 29, Day 43, Day 57)
  Cumulative incidence rates for (S)AE pattern of study participants
Individual (study participant-related) incidence of individual (S)AEs | After each of the four 14 days study episodes (Day 15, Day 29, Day 43, Day 57)
  Individual (study participant-related) incidence of individual (S)AEs
Individual (study participant-related) changes in pain severity (NRS scale) | After each of the four 14 days study episodes (Day 15, Day 29, Day 43, Day 57)
  Individual (study participant-related) changes in pain severity (measured by using 11-point numeric pain rating scale) in relation to treatment phase and loxapine dosage
Association between event pattern and individual pain level (NRS scale) | After each of the four 14 days study episodes (Day 15, Day 29, Day 43, Day 57)
  Assessment of the association between the pattern of events (Primary endpoint) related to the individual pain level (clinically relevant pain reduction is defined by an at least 30% decrease or an absolute decrease of two scale units compared to baseline using 11-point numeric pain rating scale.
Individual (study participant-related) changes in pain severity (painDETECT) | After each of the four 14 days study episodes (Day 15, Day 29, Day 43, Day 57)
  Individual (study participant-related) changes in pain severity (measured by painDETECT questionnaire) in relation to treatment phase and loxapine dosage
Association between event pattern and individual pain level (painDETECT) | After each of the four 14 days study episodes (Day 15, Day 29, Day 43, Day 57)
  Assessment of the association between the pattern of events (Primary endpoint) related to the individual changes in pain severity / characteristics measured by painDETECT questionnaire
Individual (study participant-related) changes in QoL (SF-12v2) | After each of the four 14 days study episodes (Day 15, Day 29, Day 43, Day 57)
  Individual (study participant-related) changes in the quality of life (12-item Short Form Health Survey (SF-12v2)) in relation to treatment phase and loxapine dosage
Association between event pattern and QoL (SF-12v2) | After each of the four 14 days study episodes (Day 15, Day 29, Day 43, Day 57)
  Assessment of the association between the pattern of events (Primary endpoint) related to the individual quality of life changes changes (12-item Short Form Health Survey (SF-12v2))
Individual (study participant-related) changes in anxiety and depression (HADS-D scale) | After each of the four 14 days study episodes (Day 15, Day 29, Day 43, Day 57)
  Individual (study participant-related) changes in anxiety and depression (HADS-D scale) in relation to treatment phase and loxapine dosage
Association between event pattern and anxiety and depression (HADS-D scale) | After each of the four 14 days study episodes (Day 15, Day 29, Day 43, Day 57)
  Assessment of the association between the pattern of events (Primary endpoint) related to the individual changes in anxiety and depression (HADS-D scale)
Association between event pattern and analgesic co-medication | After each of the four 14 days study episodes (Day 15, Day 29, Day 43, Day 57)
  Assessment of the association between the pattern of events (Primary endpoint) related to the individual changes in analgesic co-medication

CONTACTS AND LOCATIONS:
Overall Officials: Sven Schmiedl, MD, Study Chair — Witten/Herdecke University; Sven Schmiedl, MD, Principal Investigator — HELIOS Clinic Wuppertal
Locations (1):
- HELIOS Clinic Wuppertal, Wuppertal, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schmiedl S, Peters D, Schmalz O, Mielke A, Rossmanith T, Diop S, Piefke M, Thurmann P, Schmidtko A. Loxapine for Treatment of Patients With Refractory, Chemotherapy-Induced Neuropathic Pain: A Prematurely Terminated Pilot Study Showing Efficacy But Limited Tolerability. Front Pharmacol. 2019 Jul 25;10:838. doi: 10.3389/fphar.2019.00838. eCollection 2019. PMID 31402867